CLINICAL TRIAL: NCT05619198
Title: The Effects of Different Exercise Modalities in Adolescents With Type 1 Diabetes Using AID Systems
Acronym: MODE2022
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MODE2022
Record Dates: First submitted 2022-10-05; First posted 2022-11-16 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2022-11

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: A two-period, cross-over, clinical trial with between and within cohort comparisons of two different exercise modalities in adolescents with type 1 diabetes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Exercise (Active Comparator): Plasma and sensor glucose is monitored before, during and after a bout of high intensity interval exercise
  Interventions: Behavioral: High Intensity Interval Exercise
- Moderate Intensity Continous Exercise (Active Comparator): Plasma and sensor glucose is monitored before, during and after a bout of moderate intensity continous exercise
  Interventions: Behavioral: Moderate Intensity Continous Exercise

INTERVENTIONS:
Behavioral: High Intensity Interval Exercise — High Intensity Interval Exercise:
  * 5 minutes resting phase @ 0 watts.
  * 5-minute warm up phase @ 20 watts.
  * 40 minutes of interval work consisting of eight bouts of 1-minute cycling at a power output corresponding to ~85% of VO2max interspersed with 4-minute recovery periods at 20 watts.
  * 5 minutes resting phase @ 0 watts.
  Arms: High Intensity Interval Exercise
Behavioral: Moderate Intensity Continous Exercise — Moderate Intensity Continous Exercise:
  * 5 minutes resting phase @ 0 watts.
  * 5-minute warm up phase @ 20 watts.
  * 40 minutes of MICE 65% VO2max.
  * 5 minutes resting phase @ 0 watts.
  Arms: Moderate Intensity Continous Exercise

SUMMARY:
Objective:

The overall objective of this study is to assess the efficacy of the current recommended guidelines for physical activity (PA) in response to acute moderate intensity continous exercise (MICE) and high intensity interval exercise (HIIE) among adolescents with type 1 diabetes (T1D) using automated insulin delivery (AID) systems (MiniMed 780G and Tandem Control-IQ).

Methods:

This study will be a two-period, cross-over, clinical trial with between and within cohort comparisons of two different exercise modalities among a total of 24 age-, sex-, and insulin-dose-matched adolescents with T1D (12 using MiniMed 780G and 12 using Tandem Control-IQ).

Endpoint:

The primary endpoint is sensor-derived time in range (3.9 mmol/L-10.0 mmol/L) around exercise

DETAILED DESCRIPTION:
Participants included in the study will perform a cardiopulmonary exercise testing (CPET) before the exercise study visits, to prescribe subsequent exercise intensity thresholds. Participants will have a canula placed in a antecubital vein for plasma sampling during the test.

Participants will undertake two exercise visits each including a bout of exercise on a stationary bicycle of either one of two exercise modalities; i.) high-intensity interval exercise with sprints at ~85% of VO2max (HIIE); ii.) moderate intensity continuous exercise at ~60% of VO2max (MICE).

Participants will arrive at the research facility, Steno Diabetes Center Copenhagen, in the afternoon. As per the current recommended guidelines, the MICE-session will be announced to the AID systems 60 minutes in advance, whereas the HIIE-session will not be announced. Participants will have a canula placed in a antecubital vein for plasma sampling.

Participants will rest for 60 minutes, exercise for 45 minutes and rest again for 75 minutes before leaving the research facility. During exercise participants will be fitted with a spirometry face mask to compute ventilatory thresholds and indirect calorimetry (Vyaire Vyntus® CPX, Intramedic A/S) and a telemetry chest strap (Polar H10) for integrated HR heart rate (HR) measurements with the spirometry device.

In the MICE session: After 15 minutes post-exercise rest the temporary target/exercise mode is turned off.

Around each study visit (24 hours prior until 24 hours after), sensor glucose as well as sleep and physical activity will be recorded. Sensor glucose will be measured by participants' own devices. Sleep and physical activity level will be assessed with a wrist-worn accelerometer, ActiGraph wGT3X-BT (ActiGraph, Pensacola, FL).

Study days will be separated by at least three days.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-17 years old
* Type 1 diabetes > 1 year
* Use of Tandem t:slim X2 Control-IQ or Medtronic MiniMed 780G with connected continous glucose monitor > 3 months
* HbA1c below 75 mmol/L

Exclusion Criteria:

* Use of anti-diabetic medicine other than insulin
* Breastfeeding, pregnancy or planning to become pregnant
* Lack of compliance with key study procedures at the discretion of the investigator

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of time spent in sensor-derived time in range (3.9-10.0 mmol/L) during and after a bout of exercise | T = 0 to T = +120 (120 minutes)
  Percentage

SECONDARY OUTCOMES:
Number of hypo- (<3.9 mmol/L) and hyperglycemic (>10.0 mmol/L) occurrences during exercise session as measured by sensor and plasma sampling | T = 0 to T = +45 (45 minutes)
  Number
Percentage of time spent below (<3.9 mmol/L), in (3.9-10.0 mmol/L) and above (>10.0 mmol/L) range during in-clinic phase, measured by sensor and plasma sampling | T= -60 minutes to T= +120 minutes (3 hours)
  Percentage
Percentage of time spent below (<3.9 mmol/L), in (3.9-10.0 mmol/L) and above (>10.0 mmol/L) range during home-phase, measured by glucose sensor | 24 hours
  Percentage
Glycemic variability as coefficient of variation, measured by sensor during in-clinic phase | T= -60 minutes to T= +120 minutes (3 hours)
  Percentage
Glycemic variability as coefficient of variation, measured by plasma sampling during in-clinic phase | T= -60 minutes to T= +120 minutes (3 hours)
  Percentage
Glycemic variability as standard deviation, measured by sensor during in-clinic phase | T= -60 minutes to T= +120 minutes (3 hours)
  mmol/L
Glycemic variability as standard deviation, measured by plasma sampling during in-clinic phase | T= -60 minutes to T= +120 minutes (3 hours)
  mmol/L
Glycemic variability as coefficient of variation measured by glucose sensor during home-phase | 24 hours
  Percentage
Glycemic variability as standard deviation measured by glucose sensor during home-phase | 24 hours
  Mmol/L
Number of rescue glucose interventions to treat hypoglycemia (<3.9 mmol/L) during in-clinic and home-phase | 27 hours
  Number
Area Under the Curve and absolute concentration of serum total insulin during in-clinic phase | T= -60 minutes to T= +120 minutes (3 hours)
  Units
Dynamics of plasma glucoregulatory hormone responses during in-clinic phase | T= -60 minutes to T= +120 minutes (3 hours)
  Change in concentration
Dynamics of plasma metabolites during in-clinic phase | T= -60 minutes to T= +120 minutes (3 hours)
  Change in concentration
Glucose changes during exercise (delta change expressed as absolute [mmol/L]) during in-clinic phase | T= -60 minutes to T= +120 minutes (3 hours)
  mmol/L
Glucose changes during exercise (delta change relativized as a rate of change [mmol/min]) during in-clinic phase | T= -60 minutes to T= +120 minutes (3 hours)
  mmol/min
Amount of correction boluses given by each automated insulin delivery system during activation of temporary target and exercise mode | T= -60 minutes to T= +60 minutes (2 hours)
  Number
Comparison of heart rate (HR) during high intensity interval exercise and moderate intensity continous exercise session | T = 0 to T = +45 (45 minutes)
  Beats pr minute
Comparison of respiratory exchange ratio (RER) during high intensity interval exercise and moderate intensity continous exercise session | T = 0 to T = +45 (45 minutes)
  Ratio
Comparison of oxygen consumption (VO2) during high intensity interval exercise and moderate intensity continous exercise session | T = 0 to T = +45 (45 minutes)
  L/min
Comparison of carbon dioxide output (VCO2) during high intensity interval exercise and moderate intensity continous exercise session | T = 0 to T = +45 (45 minutes)
  L/min
Comparison of carbohydrate oxidation during high intensity interval exercise and moderate intensity continous exercise session | T = 0 to T = +45 (45 minutes)
  g/min
Comparison of lipid oxidation during high intensity interval exercise and moderate intensity continous exercise session | T = 0 to T = +45 (45 minutes)
  g/min
Comparison of resting metabolic rate after exercise session | T =+45 to T=+120 (75 minutes)
  kj/min
Plasma lactate response before, during and after cardiopulmonary exercise testing | 30 minutes
  mmol/L
Plasma glucose response before, during and after cardiopulmonary exercise testing | 30 minutes
  mmol/L
Respiratory exchange ratio (RER) collected continuously during cardiopulmonary exercise testing visit | 30 minutes
  L/min
Oxygen consumption (VO2) collected continuously during cardiopulmonary exercise testing visit | 30 minutes
  L/min
Carbon dioxide output (VCO2) collected continuously during cardiopulmonary exercise testing visit | 30 minutes
  L/min
Sleep efficiency assessed by Actigraph GT3x the night before study visits compared to after study visits. | Night 1-2
  Percentage
Wake time after sleep onset assessed by Actigraph GT3x the night before study visits compared to after study visits | Night 1- 2
  Mins
Energy expenditure assessed by Actigraph GT3x. | Day 1-3
  Kcal
Physical activity level assessed by Actigraph GT3x | Day1-3
  sedentary, light or moderate-to-vigorous

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Lindkvist, MD, Principal Investigator — Steno Diabetes Center Copenhagen, Clinical Research
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No